CLINICAL TRIAL: NCT06325852
Title: Directional Bilateral Thalamic Patterned Stimulation in Individuals with Essential Tremor
Brief Title: Directional Bilateral Thalamic Patterned Stimulation (Chronos)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alfonso Fasano (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Alfonso Fasano, MD, PhD, FAAN, Professor, University of Toronto
Organization: University of Toronto (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-5772
Record Dates: First submitted 2024-03-13; First posted 2024-03-22 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-07

CONDITIONS: Essential Tremor
Keywords: Deep Brain Stimulation; Chronos Physician Programmer
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1 (Experimental): 5 to 10 patients with tremor already treated with VIM-DBS but not doing well because of early or late loss of benefits will be recruited by the PI over a 6 months period. If interested, the potential participants will be screened, informed, and consented by a research coordinator. Before the replacement of their IPG (implantable pulse generator), a baseline measurement will be performed.
  Interventions: Other: DBS programing
- Phase 2 (Experimental): Ten patients with ET needing DBS-VIM surgery will be recruited and will receive Boston Scientific Genus IPG bilaterally connected to Boston Scientific Cartesia™ 8-contact Directional Leads. The programming will be done in four different settings/periods during the course of 8 months.
  Interventions: Other: DBS programing

INTERVENTIONS:
Other: DBS programing — The physician will utilize the Boston Scientific Chronos Clinician Programmer (software) to make adjustments to the Deep Brain Stimulation (DBS) settings for the patients.

SUMMARY:
Population Size and Eligible Patients: The investigators aim to recruit 5 to 10 patients with tremors who have previously undergone Ventral Intermedius Deep Brain Stimulation (VIM-DBS) treatment but have experienced early or late loss of benefits. Additionally, the investigators will enroll ten patients with essential tremor who require VIM-DBS surgery. These individuals will undergo bilateral implantation of Boston Scientific Genus Implantable Pulse Generator (IPG) devices, connected to Boston Scientific Cartesia™ 8-contact Directional Leads.

Study Design: This study comprises two distinct phases. Phase 1 is a cross-sectional investigation designed to identify the optimal algorithm for patterned stimulation in the VIM region . Phase 2 is a prospective clinical trial focusing on the assessment of safety and efficacy of bilateral VIM-DBS in patients with essential tremor.

Objectives: The primary objective in Phase 2 is to evaluate the safety and effectiveness of bilateral VIM-DBS in individuals with essential tremor. In Phase 1, the investigators seek to explore the impact of the Chronos programming software on tremor patients who have experienced early or late loss of benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Phase 1: 5 to 10 tremor patients already treated with VIM-DBS but not doing well due to early and/or late loss of benefits (i.e. tremor scores ON stimulation identical or greater than before surgery in absence of stimulation).
2. Phase 2: 10 Essential Tremor patients in need of DBS surgery.
3. Written and signed Informed Consent.
4. Age 18 to 85 years old.
5. Subject must have Essential Tremor, as defined by all the following criteria: (a) isolated tremor syndrome consisting of bilateral action tremor; (b) at least three years duration; and (c) with or without tremor in other locations (e.g., head, voice, or low limbs) [1].
6. Soft signs (categorizing patients as Essential Tremor-plus) will be allowed and noted in the patient's chart.
7. Subject must be on stable dose of anti-tremor medication for at least 4 weeks prior to screening.
8. Subject had no botulinum injection for at least three months prior to screening.
9. Subject does not have a significant other medical condition biasing the study finding in investigator's opinion.

Exclusion Criteria:

1. Unwilling or inability to follow the procedures specified by the protocol.
2. Presence of significant psychiatric or cognitive condition likely to compromise the subject's ability to comply with requirements of the study protocol.
3. Untreated clinically significant depression.
4. Any current drug or alcohol abuse, as determined by the investigator.
5. History of suicidal attempt within the last 1 year prior to consent or current active suicidal ideation as determined by the investigator.
6. Any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints.
7. Any terminal illness with life expectancy of < 12 months.
8. Participation in any other interventional clinical trial (e.g. drug, device).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Tremor Rating Scale (Part A-B) | Phase 1-Baseline
  Range from 0-46. with 0 representing no tremor and 46 representing severe tremor.
Tremor analysis | Phase 1-Baseline
  Using accelerometers
Tremor Rating Scale (A-C) | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  Range from 0-46. with 0 representing no tremor and 46 representing severe tremor.
Tremor analysis (meter per second squared) | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  Using accelerometers
Gait speed (meter per second) | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  Gait Analysis
Base of support (meter) | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  Gait Analysis
Step length (meter) | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  Gait Analysis
Stride length (meter) | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  Gait Analysis
Single stance time and double stance time (seconds) | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  Gait Analysis
Tandem gait | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  Gait Analysis
Posturography (newtons) | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  Using Proteokinetics Zeno System
Quality of life in Essential Tremor Questionnaire (QUEST) | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  Range from 0-40, with 0 representing no tremor and 40 representing severe tremor.
Speech analysis | Phase 2-Baseline, Month 2, Month 4, Month 6, Month 8
  automated analysis pipeline in MatLab

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorders Centre - Toronto Western Hospital, Toronto, Ontario, Canada